CLINICAL TRIAL: NCT04501848
Title: The Impact of Sleep Disordered Breathing on Parental Quality of Life
Brief Title: Parent-QoL and Sleep Disordered Breathing
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Ronen Ohad, Director Head and Neck Surgery Unit, Western Galilee Hospital-Nahariya
Other Study IDs: NHR009417
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: parents of obstructive sleep disordered breathing (OSDB) children before and after surgical treatment
  Interventions: Procedure: adenotonsillectomy
- Control: A group of parents to healthy children comprised the control group.

INTERVENTIONS:
Procedure: adenotonsillectomy — adenotonsillectomy surgery
  Groups: Study

SUMMARY:
In this prospective case-control study the investigators will enrolled parents of 45 children younger than five years of age who were planned to undergo adenotonsillectomy due to an obstructive airway indication in an academic medical center. A group of parents to healthy children will comprise the control group.

DETAILED DESCRIPTION:
Parents of children with any chronic illness may experience increased anxiety and reduced health-related quality of life (QoL).

In this study, the investigators will analyze QoL parameters among parents of obstructive sleep disordered breathing (OSDB) children before and after surgical treatment.

In this prospective case-control study the investigators will enrolled parents of 45 children younger than five years of age who are planned to undergo adenotonsillectomy due to an obstructive airway indication in an academic medical center. A group of parents to healthy children will comprisedthe control group.

The investigators will translate and validate the PAR-ENT-QoL questionnaire through forward-backward translation method.

Main outcome measure: The questionnaire was tested for reliability, consistency, reproducibility, responsiveness, and for its clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children younger than five years old who suffered from OSDB and underwent tonsillectomy or tonsillotomy with or without adenoidectomy

Exclusion Criteria:

* We excluded parents of children who required immediate surgery or had any other chronic diseases (such as ADHD, asthma, allergic rhinitis or severe medical or mental impairments).

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population included parents of children younger than five years old who suffered from OSDB and underwent tonsillectomy or tonsillotomy with or without adenoidectomy during 2018, in the Department of Otolaryngology at Galilee Medical Center, Israel.
  The control group was composed of parents of healthy children of the same age group who did not suffer from OSDB or any other acute or chronic disease and were recruited through an online survey to complete the questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
A change in the PAR-ENT-QoL questionnaire score | Change from PAR-ENT-QoL questionnaire score, 1-3 weeks before surgery to 3-9 weeks after surgery
  translated and validated the PAR-ENT-QoL questionnaire through forward-backward translation method.

CONTACTS AND LOCATIONS:
Locations (1):
- Galillee medical center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berdeaux G, Hervie C, Smajda C, Marquis P. Parental quality of life and recurrent ENT infections in their children: development of a questionnaire. Rhinitis Survey Group. Qual Life Res. 1998 Aug;7(6):501-12. doi: 10.1023/a:1008874324258. PMID 9737140
- [Background] Shteinberg YH, Eisenbach N, Sela E, Gruber M, Ronen O. Translation and cultural adaptation of the Hebrew version of the Pediatric Sleep Questionnaire: a prospective, non-randomized control trial. Sleep Breath. 2021 Mar;25(1):399-410. doi: 10.1007/s11325-020-02073-6. Epub 2020 May 12. PMID 32394315
- [Background] Koller M, Aaronson NK, Blazeby J, Bottomley A, Dewolf L, Fayers P, Johnson C, Ramage J, Scott N, West K; EORTC Quality of Life Group. Translation procedures for standardised quality of life questionnaires: The European Organisation for Research and Treatment of Cancer (EORTC) approach. Eur J Cancer. 2007 Aug;43(12):1810-20. doi: 10.1016/j.ejca.2007.05.029. Epub 2007 Aug 3. PMID 17689070
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318